CLINICAL TRIAL: NCT04265092
Title: Gaitox :Therapeutic Benefit of Incobotulinum Toxin A for Spasticity of the Triceps Surae in Patients With Multiple Sclerosis an Observational Study on Gait Spatiotemporal Parameters
Brief Title: Therapeutic Benefit of Incobotulinum Toxin A for Spasticity of the Triceps Surae in Patients With Multiple Sclerosis
Acronym: GAITOX
Status: Completed | Type: Observational
Sponsor: Pôle Saint Hélier (Other)
Responsible Party: Sponsor
Other Study IDs: Pole-sthelier
Record Dates: First submitted 2019-10-22; First posted 2020-02-11 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2019-11

CONDITIONS: Multiple Sclerosis
Keywords: Gait; Multiple Sclerosis; Spasticity; Toxin; Triceps surae
MeSH Terms: conditions — Multiple Sclerosis; Muscle Spasticity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Incobotulinum toxin A — Treatment consisted of 200 IU of incobotulinum toxinA injected into the TS. Outcome measures were assessed before injection, at 6 weeks and 3 months post-injection, using the Goal Attainment Scale (GAS), Twelve Item MS Walking (MSWS-12) Scale, Timed Up and Go (TUG) Test, 6 Minute Walk Test (6MWT). Spatiotemporal gait data was obtained by GAITRite.

SUMMARY:
Introduction/Objectives: In this observational study, we assessed the benefit following an injection of 200 international units (IU) of incobotulinum toxinA in patients with multiple sclerosis (MS) with spasticity of the triceps surae (TS) at 6 weeks (peak efficacy of toxin) and at 3 months (cancellation of efficacy).

Methods: This study enrolled all MS patients willing to participate with Expanded Disability Status Scale (EDSS) scores of less than 6, who required toxin for management of focal spasticity of the TS. Treatment consisted of 200 IU of incobotulinum toxinA injected into the TS. Outcome measures were assessed before injection, at 6 weeks and 3 months post-injection, using the Goal Attainment Scale (GAS), Twelve Item MS Walking (MSWS-12) Scale, Timed Up and Go (TUG) Test, 6 Minute Walk Test (6MWT). Spatiotemporal gait data was obtained by GAITRite.

ELIGIBILITY:
Inclusion Criteria:

* MS patients aged over 18 years
* with gait problems related to spasticity of the triceps surae,
* walking 10 m in less than a minute,
* with or without technical assistance,
* with an EDSS of 6.5 or less
* triceps surae spasticity of between 1 and 3 on the Modified Ashworth Scale.

Exclusion Criteria:

* Comprehension problems preventing the patient from expressing his/her free and informed consent to the study.
* Intolerance to botulinum toxin;
* botulinum toxin injection in the previous three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Twenty-two MS patients with a mean age of 48.2 +/- 12 years were enrolled in this study, 15 women and 7 men. In 13 patients, the disease had been in a relapsing-remitting mode for 15.2 +/- 12 years, 4 patients had secondary-progressive disease and 5 had primary progressive disease, with a mean EDSS of 4.2 +/- 1.5. Triceps surae spasticity on the Modified Ashworth Scale was 2.4 +/- 0.7.
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Spatiotemporal gait parameters | at inclusion
  Measurement of temporospatial gait parameters by GAITRite® Portable Gait Analysis Walkway: gait velocity (m/sec)
Spatiotemporal gait parameters | at inclusion
  Measurement of temporospatial gait parameters by GAITRite® Portable Gait Analysis Walkway: cadence (nb/sec)
Spatiotemporal gait parameters | at inclusion
  Measurement of temporospatial gait parameters by GAITRite® Portable Gait Analysis Walkway: duration of stance time on the injected and non-injected side (in sec)
Spatiotemporal gait parameters | at inclusion
  Measurement of temporospatial gait parameters by GAITRite® Portable Gait Analysis Walkway: duration of swing time on the injected and non-injected side (in sec)
Spatiotemporal gait parameters | at inclusion
  Measurement of temporospatial gait parameters by GAITRite® Portable Gait Analysis Walkway: step length on the injected and non-injected side (in meters)
Spatiotemporal gait parameters | at inclusion
  Measurement of temporospatial gait parameters by GAITRite® Portable Gait Analysis Walkway: support distribution (in %).
Spatiotemporal gait parameters | At six weeks
  Measurement of temporospatial gait parameters by GAITRite® Portable Gait Analysis Walkway: gait velocity (m/sec)
Spatiotemporal gait parameters | At six weeks
  Measurement of temporospatial gait parameters by GAITRite® Portable Gait Analysis Walkway: cadence (nb/sec)
Spatiotemporal gait parameters | At six weeks
  Measurement of temporospatial gait parameters by GAITRite® Portable Gait Analysis Walkway: duration of stance time on the injected and non-injected side (in sec)
Spatiotemporal gait parameters | At six weeks
  Measurement of temporospatial gait parameters by GAITRite® Portable Gait Analysis Walkway: duration of swing time on the injected and non-injected side (in sec)
Spatiotemporal gait parameters | At six weeks
  Measurement of temporospatial gait parameters by GAITRite® Portable Gait Analysis Walkway: step length on the injected and non-injected side (in meters)
Spatiotemporal gait parameters | At six weeks
  Measurement of temporospatial gait parameters by GAITRite® Portable Gait Analysis Walkway: support distribution (in %).
Spatiotemporal gait parameters | At three months
  Measurement of temporospatial gait parameters by GAITRite® Portable Gait Analysis Walkway: gait velocity (m/sec)
Spatiotemporal gait parameters | At three months
  Measurement of temporospatial gait parameters by GAITRite® Portable Gait Analysis Walkway: cadence (nb/sec)
Spatiotemporal gait parameters | At three months
  Measurement of temporospatial gait parameters by GAITRite® Portable Gait Analysis Walkway: duration of stance time on the injected and non-injected side (in sec)
Spatiotemporal gait parameters | At three months
  Measurement of temporospatial gait parameters by GAITRite® Portable Gait Analysis Walkway: duration of swing time on the injected and non-injected side (in sec)
Spatiotemporal gait parameters | At three months
  Measurement of temporospatial gait parameters by GAITRite® Portable Gait Analysis Walkway: step length on the injected and non-injected side (in meters)
Spatiotemporal gait parameters | At three months
  Measurement of temporospatial gait parameters by GAITRite® Portable Gait Analysis Walkway: support distribution (in %).

SECONDARY OUTCOMES:
Six-Minute Walk Test (6MWT) | at inclusion, at 6 weeks, at three months
  The 6 MWT is a simple test which requires a 30-meter course, calm, indoors, flat, in a rectilinear rectangular corridor. The route is marked every 3 meters with colored marks. The U-turn should be viewed with a cone. The purpose of this test is to walk as much as possible for 6 minutes. The score is between 0 meters for a non-ambulatory person and about 900 meters for a healthy subject.
the Multiple Sclerosis Walking Scale (MSWS-12) | at inclusion, at 6 weeks, at three months
  From the numbers circled against these questions, the healthcare professional can calculate the MSWS-12 score. This is done by adding the numbers you have circled, giving a total out of 60, and then transforming this to a scale with a range from 0 to 100. Higher scores indicate a greater impact on walking than lower scores.
the Goal Attainment Scale (GAS) score with determination | at inclusion, at 6 weeks, at three months
  In collaboration with the patient, the doctor define a primary and a secondary objectives, with a specific mark for each: -2: worse than before, -1: no change, 0: objective achieved, 1: result better than expected, 2: unexpected result
The Timed Up and Go test (TUG) | at inclusion, at 6 weeks, at three months
  TUG performance is rated on a scale of 1 to 5, where 1 indicates "normal functioning" and 5 indicates "severe abnormal behavior", according to the individual's perception of the risk of falling (Podsiadlo & Richardson, 1991) . The score consists of the time taken to complete the test, in seconds.

IPD SHARING:
Plan to Share IPD: No
This prospective study is an observational pilot study, which seeks to evaluate the impact of a common treatment, as administered on a daily basis, without any change in the patients usual treatment pathway.